CLINICAL TRIAL: NCT02559115
Title: A Phase II Study of 68Ga-RM2 for PET/CT of Gastrin Releasing Peptide Receptor (GRPr) Expression in Prostate Cancer
Brief Title: 68Ga-RM2 for PET/CT of Gastrin Releasing Peptide Receptor (GRPr) Expression in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-146
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2020-06

CONDITIONS: Prostate Cancer
Keywords: 68Ga-RM2; PET/CT scan; Gastrin Releasing Peptide Receptor (GRPr); 14-146
MeSH Terms: conditions — Prostatic Neoplasms | interventions — BAY 86-7548; Positron Emission Tomography Computed Tomography

ARMS (1):
- PET/CT imaging with 68Ga-RM2 (Experimental): The intervention is the administration of a single dose of 150-200 MBq 68Ga-RM2 (mass <= 30 μg) for imaging purposes. This will be followed by a 30-40 min PET/CT study after a waiting period of 60 min (+/- 10 min). Prior clinical experience suggests that imaging can be performed within 1 hour post injection (27, 28). MR imaging and prostatectomy will be performed as standard of care at MSKCC.
  Interventions: Radiation: 68Ga-RM2 (RM2); Device: PET/CT Scan

INTERVENTIONS:
Radiation: 68Ga-RM2 (RM2)
Device: PET/CT Scan

SUMMARY:
The purpose of this study is to see if a new diagnostic research agent named 68Ga-RM2 can show prostate cancer on a PET/CT scan. 68Ga-RM2 stands for Galium-68 labeled DOTA-4-amino-1-carboxymethylpiperidine-D-Phe-Gln-Trp-Ala-Val-Gly-His-Sta-Leu-NH2. This study is being done because there are unmet medical needs to improve the current ways of detecting prostate cancers before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Biopsy proven adenocarcinoma of the prostate
* Patients with low-risk, intermediate-risk and high-risk tumors according to NCCN guidelines (2.2014) will be included
* Planned radical prostatectomy at MSKCC
* Multiparametric MRI of the pelvis (performed or planned) as routine care

Exclusion Criteria:

* Patients meeting any of the following exclusion criteria will not be eligible for study entry:
* Hematologic

  * Platelets <75K/mcL
  * ANC <1.0 K/mcL
* Hepatic laboratory values

  * Bilirubin >2.0 x ULN (institutional upper limits of normal)
  * AST/ALT >2.5 x ULN
* Renal laboratory values

  o Creatinine > 2.0 x ULN
* Claustrophobia interfering with MRI and PET/CT imaging
* Prior pelvic radiation
* Prior androgen deprivation therapy
* Patients deemed not surgical candidates due to prohibitive co-morbidities

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Vargas Alvarez, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- PET/CT Imaging With 68Ga-RM2: The intervention is the administration of a single dose of 150-200 MBq 68Ga-RM2 (mass <= 30 μg) for imaging purposes. This will be followed by a 30-40 min PET/CT study after a waiting period of 60 min (+/- 10 min). Prior clinical experience suggests that imaging can be performed within 1 hour post injection (27, 28). MR imaging and prostatectomy will be performed as standard of care at MSKCC.
  68Ga-RM2 (RM2)
  PET/CT Scan
Period: Overall Study
Arm/Group | PET/CT Imaging With 68Ga-RM2
Started | 19
Completed | 16
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | PET/CT Imaging With 68Ga-RM2
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 60 [45 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Localizing Tumors
Description: Localization will be defined using a total of 12 regions within the prostate: right and left base, midgland and apex in both peripheral and transition zones. The uptake on each region will be assessed by a radiologist blinded to standard of care imaging and clinical characteristics. Histopathological confirmation will be used as the gold standard.
Time Frame: within two weeks prior to the planned prostatectomy
Measure: Number; unit: Areas of the body
Units Other Than Participants: Areas Analyzed
Arm/Group | PET/CT Imaging With 68Ga-RM2
Number analyzed (Participants) | 19
Number analyzed (Areas Analyzed) | 192
Areas of the body
  Containing cancer | 128
  Not containing cancer | 64

ADVERSE EVENTS:
Time Frame: Up to 1 day following study intervention.
Arm/Group | PET/CT Imaging With 68Ga-RM2
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 6/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PET/CT Imaging With 68Ga-RM2 (N=19)
Lymphocyte count decreased (Investigations) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/15/NCT02559115/Prot_SAP_000.pdf